CLINICAL TRIAL: NCT03172403
Title: Skeletal Muscle Expression of Myostatin and Cancer of Digestive System Associated Cachexia(MYOCAC Study)
Brief Title: Skeletal Muscle Expression of Myostatin and Cancer of Digestive System Associated Cachexia
Acronym: MYOCAC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped prematurely by decision of the sponsor due to lack of inclusion.
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1708054; ANSM (Other: 2017-A01233-50)
Record Dates: First submitted 2017-05-23; First posted 2017-06-01 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Cancer of Digestive System
Keywords: Cachexia; Cancer of Digestive System; Myostatin; Skeletal muscle
MeSH Terms: conditions — Digestive System Neoplasms; Cachexia | interventions — Body Height; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with digestive cancer requiring resection surgery (Experimental): Patients with cancer of digestive system requiring resection surgery will be included. They will have measure of height and weight, blood samples, skeletal muscle force, skeletal muscle index and muscle biopsy.
  V1: Inclusion will be effectuated at the time of anaesthetic consultation V2: The day before and day of resection surgery about 1 month after V3: Follow-up at 1 month V4: Follow-up at 3 months V6: Follow-up at 6 months
  Interventions: Diagnostic Test: Height and weight; Diagnostic Test: Blood samples; Diagnostic Test: Skeletal muscle force; Diagnostic Test: Skeletal muscle index; Diagnostic Test: Muscle biopsy

INTERVENTIONS:
Diagnostic Test: Height and weight — Height and weight will be measured to estimate cachexia degree at the time of anaesthetic consultation. (V1)
Diagnostic Test: Blood samples — Blood samples will be collected for measuring myostatin on blood at the time of anaesthetic consultation, the day before resection surgery, follow-ups at 1, 3 and 6 months. (V1, V2, V3, V4, V6)
Diagnostic Test: Skeletal muscle force — Skeletal muscle force will be determined from Computerized Tomography (CT)-scan at the time of anaesthetic, follow-ups at 1, 3 and 6 months. (V1, V3, V4, V6)
Diagnostic Test: Skeletal muscle index — Skeletal muscle index will be determined from Computerized Tomography (CT)-scan at the time of anaesthetic, follow-ups at 1, 3 and 6 months. (V1, V3, V4, V6)
Diagnostic Test: Muscle biopsy — Muscle biopsy will be performed during resection surgery under general anaesthesia. (V2)

SUMMARY:
Cancer cachexia is responsible for the death of approximately 20% of patients. Myostatin is a master negative regulator of skeletal muscle mass. If the role of myostatin in cancer cachexia is now well established in murine models, no study has focused on muscle expression of Myostatin in relation to the degree of cachexia. the hypothesize is that muscle Myostatin a biological marker of cachexia in patients with cancer of digestive system. The main objective is to compare skeletal muscle Myostatin messenger RiboNucleic Acid (mRNA) level as a function of cachexia in cancer of digestive system patients. Myostatin messenger RiboNucleic Acid (mRNA) level will be determined in a muscle sample taken during the resection under general anaesthesia. Skeletal muscle index will be determined before surgery, 3 and 6 months after surgery. Muscle strength of the lower and upper limbs will be determined before resection, at 1 month, 3 months and 6 months postoperatively. Blood sampling will also be performed on these 4 occasions.

ELIGIBILITY:
Inclusion Criteria:

* Women and men aged 40-80.
* Diagnosis for cancer of digestive system requiring surgery with neoadjuvant treatment or not.
* Signature of consent
* Affiliate or beneficiary of social security

Exclusion Criteria:

* Administration of corticosteroids.
* Thyroid disease treated.
* Severe chronic pathology during treatment (neuro-muscular pathologies, renal insufficiency requiring dialysis, COPD under continuous oxygen therapy).
* Psychological, familial, social or geographical conditions that could affect the participation of the subject throughout the duration of the protocol.
* BMI> 30 due to the difficulty of interpretation of BMI variations in obese patients

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2019-01-03 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Correlation between skeletal muscle and degree myostatin | Day 1
  Evaluate correlation between skeletal muscle force/index and degree myostatin. Skeletal muscle force/index will be determinated by skeletal muscle force/index results.
  Degree myostatin will be determinated by blood samples with Enzyme Linked ImmunoSorbent Assay (ELISA) method.

SECONDARY OUTCOMES:
Correlation between skeletal muscle force and index before resection surgery | Baseline from 7 months
  Evaluate Correlation between skeletal muscle force and index before resection surgery to estimate the extent of cachexia-induced muscle dysfunction by results tests.
Correlation between level of myostatin muscular expression and degree myostatin | Month 2
  Evaluate correlation between level of myostatin muscular expression and degree myostatin.
  Level of myostatin muscular expression will be determinated by muscle biopsy. Degree myostatin will be determinated by blood samples with Enzyme Linked ImmunoSorbent Assay (ELISA) method.
Correlation between level of myostatin muscular expression and skeletal muscle force and index after resection surgery | Month 2
  Determinate correlation between level of myostatin muscular expression and skeletal muscle force and index after resection surgery.
Correlation between level of myostatin muscular expression and skeletal muscle force and index after resection surgery | Month 4
  Determinate correlation between level of myostatin muscular expression and skeletal muscle force and index after resection surgery.
Correlation between level of myostatin muscular expression and skeletal muscle force and index after resection surgery | Month 7
  Determinate correlation between level of myostatin muscular expression and skeletal muscle force and index after resection surgery.
Analysis level of myostatin muscular expression and blood samples results | Month 2
  Analysis level of myostatin muscular expression and blood samples results according to cancer stage, neoadjuvant treatment and chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Karine ABBOUD, MD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No